CLINICAL TRIAL: NCT02746172
Title: Clinical Metrics for Assessing Audibility, Comfort and Performance of Cochlear Implant Recipient MAPs
Brief Title: Clinical Metrics for Assessing Cochlear Implant Recipient MAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Royal Victoria Eye and Ear Hospital (Other Government); Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC5628
Record Dates: First submitted 2016-04-13; First posted 2016-04-21 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: cochlear implants; Mapping; in-situ audiometry
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cochlear Implant Recipients (Experimental): cochlear implant recipients
  Interventions: Device: Cochlear implant with in-situ audiometry
- Normal Hearing Volunteers (No Intervention): Normal hearing volunteers

INTERVENTIONS:
Device: Cochlear implant with in-situ audiometry
  Arms: Cochlear Implant Recipients

SUMMARY:
The aim of this research is to investigate the potential use of specific metrics in assessing the quality and optimising an individual's cochlear implant fitting. Assessment of the sensitivity and specificity of specific metrics that are potential predictors of inaccurate T-levels and C-levels is important to determining best methods for streamlined high quality fitting, providing the potential for feedback to the individual and clinic, as well as automated adjustments for optimisation. Ultimately the objective is to increase clinical capacity for managing both the installed base and new candidates for cochlear implantation.

DETAILED DESCRIPTION:
Optimising the clinical fitting of a cochlear implant to an individual listener is an important aspect of post-operative clinical care. The level of success experienced by any individual with a cochlear implant can be influenced, to a significant extent, by the quality of the clinical programming by the audiologist. During clinical programming the audiologist typically measures the amount of electrical charge required to elicit first hearing (the T-level) and to provide a loud but comfortable percept (the C-level) on each of the 22 electrodes. The amount of electrical stimulation required for a threshold and a comfortably loud percept varies across the electrodes of the array and also across individual users. Appropriately set lower and upper electrical stimulation levels are vital for ensuring that the listener is able to detect reasonably soft sounds whilst loud sounds are perceived as loud while remaining comfortable. Achieving this result across the relevant frequency range is a prime aim of programming.

There are a number of challenges in achieving optimal fitting of cochlear implant recipients in the clinical setting. First, there are varying skill levels and experience level of health professionals and allied workers involved in programming devices for cochlear implant recipients, often resulting in variability in the quality of the program (or MAP) provided to an individual. Second, there are varying levels of access to specialized equipment such as sound booths which are required for some types of audiometric measures to be reliably obtained. Finally, there are increasing demands on clinical capacity, with the specialized centres typically treating recipients having limited resources and ability to effectively manage the rapidly increasing population.

As a result, there is an increased need for effective, quality-controlled but streamlined management of implanted recipients.

The aim of the current study is to investigate the potential use of specific metrics in assessing the quality and optimizing an individual's cochlear implant fitting. Assessment of the sensitivity and specificity of specific metrics that are potential predictors of inaccurate T-levels and C-levels is important to determining best methods for streamlined high quality fitting, as well as automated adjustments for optimizing. One of the key objectives is to integrate a new technological advance in the form of in-situ audiometry, which removes the need for a sound booth to conduct audibility checks of the program. Other planned investigations relate to identifying the metrics which best identify maps that are not optimized, and to development and assessment of a range of techniques which may be able to be effectively applied in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years) cochlear implant recipients
2. Implanted with the CI500, CI24RE and Nucleus 24 Series and CI422 cochlear implants.
3. User of commercially available Freedom, CP810 or CP900 series sound processor
4. User of the ACE strategy
5. At least 3 months experience with the cochlear implant
6. Fluent speaker in the language used to assess speech perception performance
7. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Additional handicaps that would prevent participation in evaluations
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Sensitivity of percentage words/ phonemes correct, in detecting MAPs with inaccurate T and C levels in cochlear implant MAPs. | Testing over 12 weeks
Sensitivity of speech reception threshold for numbers and sentences in noise, in detecting MAPs with inaccurate T and C levels in cochlear implant MAPs. | Testing over 12 weeks
Sensitivity of aided hearing thresholds, in detecting MAPs with inaccurate T and C levels in cochlear implant MAPs. | Testing over 12 weeks
Sensitivity of loudness ratings for narrow band noise presented at different frequencies and levels, in detecting MAPs with inaccurate T and C levels in cochlear implant MAPs. | Testing over 12 weeks

SECONDARY OUTCOMES:
Test-retest reliability of in-situ aided audiometry | Testing over 6 weeks
  This will be compared to the test-retest reliability of free-field aided audiometry which is within a margin of 10 dB HL.

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No